CLINICAL TRIAL: NCT05460819
Title: A Randomized Controlled Trial Study of Acupuncture in the Treatment of Hot Flashes in Patients With Hormone Receptor-positive Breast Cancer.
Brief Title: Acupuncture for Hot Flashes in Patients With Hormone Receptor-positive Breast Cancer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Qianyan Liu, Principal Investgator, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022JC-55
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hot Flashes; Breast Cancer; Acupuncture
Keywords: breast cancer; Acupuncture; hot flashes; Functional MRI
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): Treatment group A was given endocrine and acupuncture treatment for 8 weeks (24 times in total, 3 times a week); followed up for 16 weeks, no acupuncture treatment.
  Interventions: Other: Acupuncture treatment
- Treatment group B (Sham Comparator): Treatment group B was given endocrine and sham acupuncture treatment for 8 weeks, followed up for 16 weeks, no acupuncture during the period, and after 16 weeks, received standardized acupuncture for 8 weeks (24 times in total, 3 times a week).
  Interventions: Other: Sham Acupuncture treatment
- control (No Intervention): The control group was given conventional adjuvant endocrine therapy, premenopausal patients received tamoxifen therapy, and postmenopausal patients received aromatase inhibitor or tamoxifen therapy.

INTERVENTIONS:
Other: Acupuncture treatment — Acupoint selection: Hegu-Yinxi acupoint group (clearing heat and relieving sweat), Sanyinjiao-Fuliu acupoint group (nourishing yin and tonifying kidney), Tianshu-uteri acupoint group (special effect points) (12 acupoints on both sides).
  Frequency: 3 times a week (once every other day) for a total of 8 weeks of continuous treatment.
  Operation: Use a one-time sterile acupuncture needle (0.30×40mm, Huatuo brand), insert the needle 0.5 inch along the anatomical position, level up and relieve the qi, and keep the needle for 20 minutes.
  Arms: Treatment group A
Other: Sham Acupuncture treatment — Selecting acupoints: Select the side opening positions of the 6 acupuncture points in the real acupuncture group, and select non-meridian and non-points (points with less nerve distribution, sparseness, and rich muscles).
  Frequency: 3 times a week (once every other day) for a total of 8 weeks of continuous treatment.
  Operation: ① Shallow needling scheme: use a disposable sterile acupuncture needle, insert the needle 0.2 inch, without twisting, and keep the needle for 20 minutes. ②Non-invasive acupuncture plan: choose a special comfort needle with no needle tip at the top of the needle, paste a disposable sterile foam pad on the non-acupoint, and use a disposable sterile flat head The acupuncture needles were pierced into the foam pad, lightly touching but not piercing the skin, and not breathing; the needles were kept for 20 minutes.
  Arms: Treatment group B

SUMMARY:
This study intends to further evaluate the efficacy of acupuncture by comparing the intervention effects of different acupuncture treatment regimens on hot flashes in breast cancer ; and to explore the central effect regulation mechanism of acupuncture intervention on hot flashes based on functional magnetic resonance imaging technology.

DETAILED DESCRIPTION:
This topic combines the theory of "unblocking the governor and warming the yang" with the important findings of modern research, that is, the important mechanism of the spine in the pathogenesis of breast cancer, and innovatively proposes the technique of unblocking the governor and treating the spine. Prospective clinical intervention research in rehabilitation, objectively evaluate the clinical efficacy, advantages and disadvantages of this technology, so as to effectively break through the current application dilemma of acupuncture and bone-setting manipulation in tumor diseases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old;
* Adjuvant hormone therapy (eg, tamoxifen and/or aromatase inhibitors) with or without ovarian function suppression has been administered for at least 4 weeks and is currently on treatment;
* Vasomotor syndrome for at least 6 weeks;
* Premenopausal or postmenopausal patients;
* Patients with persistent hot flashes for at least 4 weeks and with a frequency of more than 14 hot flashes per week (2 times per day) in the week before inclusion in the study, the weekly average hot flash composite score is 3-4;
* Patients after surgery and after chemotherapy (if any);
* Eastern Cooperative Oncology Group score of 0-1 points.
* Sign the informed consent and voluntarily participate in this clinical observation.

Exclusion Criteria:

* Tumor metastases, undergoing chemoradiotherapy or planning surgery;
* Pharmacological intervention for hot flashes with hot flash treatment drugs such as selective serotonin reuptake inhibitors (SSRIs) and/or anticonvulsants for at least 4 weeks prior to study initiation;
* Unstable heart disease or myocardial infarction within 6 months prior to study start;
* Started or changed adjuvant hormone therapy within the past week, or who planned to start or change adjuvant hormone therapy in the past 14 weeks;
* Seizures of unknown likelihood or history of seizures;
* Have used acupuncture for hot flashes within 6 months prior to the start of the study;
* Pregnant or breastfeeding patients;
* Apparent uncontrolled infection;
* Mental illness or family history; neurological disorder or family history.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in cancer therapy functional assessment | Baseline, 8,24 weeks later
  Cancer therapy functional assessment scores will be assessed with Cancer Therapy Functional Assessment-Breast cancer, version 4.The minimum value is 0 , and the maximum value is 185. The higher scores mean a worse outcome.
Change in acupuncture efficacy expectation assessment | Baseline, 8,24 weeks later
  Acupuncture efficacy expectation assessment scores will be assessed with acupuncture efficacy expectation assessment. The minimum value is 0 , and the maximum value is 20. The higher scores mean a better outcome.
Change of functional connectivity of whole brain | Baseline, 8,24 weeks later
  Functional connectivity will be measured with magnetic resonance imaging based on blood oxygen level dependence.
Change of metabolism of glucose in the brain | Baseline, 8,24 weeks later
  Accumulation of 18F-fluorodeoxyglucose(18F-FDG) will be analyzed by time-related Positron emission tomography.
Change of hot flash severity | Baseline, 8,24 weeks later
  Hot flash severity will be assessed with hot flash scores each week. There are four levels of severity： Mild: Duration: Less than five minutes. Symptoms: warmth, discomfort, flushing. Moderate: Duration: Up to fifteen minutes. Symptoms: warmth in head, neck, ears, or body; tense, tight muscles; clammy skin; change in heart rate or rhythm; light sweating; dry mouth.
  Severe: Duration: Up to twenty minutes. Symptoms: Fever, sometimes like a crucible or burning sensation; change in heart rate or rhythm; feeling faint; headache; heavy sweating.
  Very severe: Duration: Up to forty-five minutes. Symptoms: boiling heat; constant sweating; trouble breathing; feeling faint, dizzy; leg cramps or feeling cramps; change in heart rate; stomach upset.
  The greater severity mean a worse outcome.

SECONDARY OUTCOMES:
Change in sleep | Baseline, 8,24 weeks later
  Sleep scores will be assessed with Pittsburgh sleep quality index.The minimum value is 9, and the maximum value is 36. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Bai, phd, Study Director — Xi'an Jiaotong University
Locations (1):
- Jiangsu Province Hospital of Traditional Chinese Medcine, Nanjing, Jiangsu, China